CLINICAL TRIAL: NCT03637920
Title: Sexuality in Transmen During Hormone and Operative Treatment Compared to Cisgender Women and Men: a Follow-up Study
Brief Title: Sexuality in Transmen During Hormone and Operative Treatment
Acronym: Transmann
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 30-087 ex 17/18
Record Dates: First submitted 2018-08-10; First posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Gender Dysphoria; Gender Identity Disorder; Transsexualism; Body Image; Sexuality
Keywords: Transmen; Sexuality; Sexual behavior; Body Image; Trassexualism
MeSH Terms: conditions — Gender Dysphoria; Transsexualism; Sexuality; Sexual Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- transmen: Biological women, who identify as men and are seeking gender reassignment.

SUMMARY:
With this analysis the investigators aim at discovering a difference in sexuality between transmen, cissexual women and cissexual men. A potential impact of body satisfaction will also be explored. Furthermore the investigators want to assess the gender dysphoria in transmen.

DETAILED DESCRIPTION:
The aim of the study is to investigate transmen's sexuality and body satisfaction during hormonal and surgical reassignment. Furthermore sexual orientation, sexual behavior and gender dysphoria will be assessed.

Therefore an online survey with five measurements throughout the gender reassignment treatment is conducted. As a matter of Routine, postoperative complications will be recorded retrospectively. To compare transmen's data with cisgender women and men we will be using data of the questionnaire's validation studies.

The following questionnaires are used:

Sexuality: Multidimensionaler Fragebogen zur Sexualität (Brenk-Franz & Strauß, 2011).

Sexual orientation: Fragebogen zur Sexualgeschichte und zum sexuellen Verhalten (Brenk, 2005) Gender dysphoria: Utrecht Gender Dysphoria Scale (Cohen-Kettenis & Van Goozen, 1997) Body image: Fragebogen zum Körperbild (Clement & Löwe, 1996) Sociodemographic questionnaire: age, education, work, living situation, relationship status, gender reassignment treatment so far, coming out Case report form

T0: baseline measurement (patient is at the start of the hormonal treatment or has already startet but has not undergone any gender reassignment surgery) T1: within 2 weeks before the mastectomy T2: 6 months (+/- 2 weeks) after mastectomy T3: 6 months (+/- 2 weeks) after colpectomy T4: 6 months (+/- 2 weeks) after the last gender reassignment surgery

ELIGIBILITY:
Inclusion Criteria:

* Transsexualism (Female to Male) approved by a psychologist's oder psychiatrist's report
* good German skills
* fully competent
* good computer skills

Exclusion Criteria:

* insufficient German
* patient rejects the participation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The study includes persons who were born as women, but identify as men.
Study Population: The study includes biological women, who identify as men and are planning to go through gender reassignment. The participants age is between 18 and 50.
  Participants are recruited at the Medical University Hospital of Graz and the consulting center "Courage".
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2018-07-30 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Changes in sexuality due to hormonal treatment using the Multidimensional Sexuality Questionnaire | 2 years
  The Multidimensional Sexuality Questionnaire (German version: Multidimensionaler Fragebogen zur Sexualität; Brenk-Franz & Strauß, 2011) assesses 12 different aspects of sexuality and consists of 60 items on a scale from 1 to 5. It also includes one nominal item, which refers to the relationship status. Sum scores are formed for each subscale (high scores indicate high value).

SECONDARY OUTCOMES:
Changes in sexuality due to surgical reassignment using the Multidimensional Sexuality Questionnaire | 5 years
  The Multidimensional Sexuality Questionnaire (German version: Multidimensionaler Fragebogen zur Sexualität; Brenk-Franz & Strauß, 2011) assesses 12 different aspects of sexuality and consists of 60 items on a scale from 1 to 5. It also includes one nominal item, which refers to the relationship status. Sum scores are formed for each subscale (high scores indicate high value).
Changes in sexual history due to surgical reassignment using the Fragebogen zur Sexualgeschichte und zum sexuellen Verhalten | 5 years
  The Fragebogen zur Sexualgeschichte und zum sexuellen Verhalten (Brenk, 2005) is a 16-item scale, with various answer schemes on sexual behavior and sexual history.
Changes in body image during sexual reassignment therapy using the Fragebogen zum Körperbild | 5 years
  Body image will be measured with the Fragebogen zum Körperbild (Clement & Löwe, 1996) including 20 items on a scale of 1-5. 10 Items measure negative body assessment (min. 10, max. 50) and the other 10 items measure vital body dynamic (min. 10, max. 50); sum scores are formed for both scales, in which high scores represent high values in each scale.
Gender dysphoria using the Utrecht Gender Dysphoria Scale | 5 years
  The Utrecht Gender Dysphoria Scale (Cohen-Kettenis & Van Goozen, 1997) is a 12-item questionnaire and is the primary measure used to assess gender dysphoria. Each item is scored on a scale from 1 to 5 and a sum score is calculated with a min. of 12 and a max. of 60 (high sum scores represents a more severe gender dysphoria).
Sexuality in transmen compared to cisgender women and men using the Multidimensional Sexuality Questionnaire | 5 years
  The Multidimensional Sexuality Questionnaire (German version: Multidimensionaler Fragebogen zur Sexualität; Brenk-Franz & Strauß, 2011) assesses 12 different aspects of sexuality and consists of 60 items on a scale from 1 to 5. It also includes one nominal item, which refers to the relationship status. Sum scores are formed for each subscale (high scores indicate high value).
Sexual history in transmen compared to cisgender women and men using the Fragebogen zur Sexualgeschichte und zum sexuellen Verhalten | 5 years
  The Fragebogen zur Sexualgeschichte und zum sexuellen Verhalten (Brenk, 2005) is a 16-item scale, with various answer schemes on sexual behavior and sexual history.
Changes in sexual history due to hormonal treatment using the Fragebogen zur Sexualgeschichte und zum sexuellen Verhalten | 2 years
  The Fragebogen zur Sexualgeschichte und zum sexuellen Verhalten (Brenk, 2005) is a 16-item scale, with various answer schemes on sexual behavior and sexual history.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Ulrich, Assoc Prof, MD PhD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University Graz, Graz, Styria, Austria